CLINICAL TRIAL: NCT03839160
Title: The Efficacy of Serratus Anterior Plane Block in Analgesia for Thoracotomy: a Prospective Study
Brief Title: The Efficacy of Serratus Anterior Plane Block (ESAPB) for Thoracotomy: a Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: truncal block SAPB
Record Dates: First submitted 2017-11-23; First posted 2019-02-15 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Pain, Postoperative; Anesthesia; Thoracotomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAPB group. Group S (Active Comparator): In this group, serratus anterior plane block (SAPB) was performed before extubation with injection of 30 ml of 0.25% bupivacaine hydrochloride followed by 0.1ml/kg/hr of 0.12% bupivacaine hydrochloride. In addition to SAPB, intravenous patient-controlled-analgesia morphine was used. Morphine solution was prepared at a concentration of 0.5 mg/mL with the device programmed to 2 mg of bolus dose and 10 min of locking time.
  Interventions: Procedure: Serratus anterior plane block; Drug: Intravenous patient-controlled-analgesia morphine
- Control group. Group C (Placebo Comparator): In this group, intravenous patient-controlled-analgesia morphine was used. Morphine solution was prepared at a concentration of 0.5 mg/mL with the device programmed to 2 mg of bolus dose and 10 min of locking time.
  Interventions: Drug: Intravenous patient-controlled-analgesia morphine

INTERVENTIONS:
Procedure: Serratus anterior plane block — Serratus anterior plane block was applied in Group S. It was performed at the end of the operation following the skin closure, while the patient lay on his side with his arm above the head. After proper site cleaning, the first and second ribs were identified with a linear probe in the midclavicular line. The USG probe was advanced caudally in the sagittal plane, and the fourth and fifth ribs were visualized. The USG probe was then directed posteriorly and the serratus, latissimus dorsi and intercostal muscles were visualized. Bupivacaine 0.25% 30 mL was administered to the lower plane of the serratus muscle through an inserted catheter under the guidance of USG through the in-line technique. Afterwards, 0.12% bupivacaine hydrochloride was maintained at the rate of 0.1ml/kg/hr.
  Other Names: Serratus plane block
  Arms: SAPB group. Group S
Drug: Intravenous patient-controlled-analgesia morphine — Morphine solution was prepared at a concentration of 0.5 mg/mL with the device programmed to 2 mg of bolus dose and 10 min of locking time.
  Other Names: PCIA

SUMMARY:
Thoracotomy is considered the most painful surgical procedure. Ultrasound-guided serratus anterior plane block (SAPB) is a relatively new truncal block method treating thoracotomy pain. In this study, investigators aim to ascertain the efficacy of SAPB in thoracotomy.

DETAILED DESCRIPTION:
Thoracotomy is considered the most painful surgical procedure, even with thoracic epidural analgesia (TEA) as a golden standard for acute post-thoracotomy pain. Ultrasound-guided serratus anterior plane block (SAPB) is a relatively new truncal block method treating thoracotomy pain, yet more evidence is needed to ascertain its efficacy.

This is a prospective study carried out in a tertiary hospital. Patients scheduled for thoracotomy are randomized into two groups: Group M (intravenous patient-controlled-analgesia morphine) and Group S (intravenous patient-controlled analgesia morphine and SAPB). Morphine consumption, VAS pain score and Prince-Henry pain score are recorded for 72 hours respectively at PACU, 2hr, 6hr, 12hr, 24hr, 48hr and 72hr, with heart rate, systolic pressure, diastolic pressure, mean arterial pressure and SpO2. Moreover, the profile of opioids-related side effects and length of hospital stay are documented. The primary objective of the study is to evaluate the efficacy of SAPB. The secondary objective is to compare the opioids-related side effects (including nausea, vomiting and pruritus), hemodynamic parameters and the length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* BMI 18-28kg/m2
* Wedge incision and lobectomy

Exclusion Criteria:

* Uncontrolled hypertension or chronic conditions
* History of opioid dependence
* Allergy to bupivacaine hydrochloride
* Severe bleeding during operation or post operation
* Inability to communicate with investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale | Changes at 2hr, 6hr, 12hr, 24hr, 48hr and 72hr post-operation
  Adult Pain Visual Analog Scale

SECONDARY OUTCOMES:
Hemodynamic profile - Heart rate | At 2hr, 6hr, 12hr, 24hr, 48hr and 72hr post-operation
  Heart rate
Hemodynamic profile - blood pressure | At 2hr, 6hr, 12hr, 24hr, 48hr and 72hr post-operation
  blood pressure
Hemodynamic profile - SpO2 | At 2hr, 6hr, 12hr, 24hr, 48hr and 72hr post-operation
  SpO2
Opioids-related side effects - nausea | At 2hr, 6hr, 12hr, 24hr, 48hr and 72hr post-operation
  nausea
Catheter-related profile | at Day 1, Day2 and Day 3 post-operation
  The position of the catheter tip and the level of blockade
Morphine consumption | At 2hr, 6hr, 12hr, 24hr, 48hr and 72hr post-operation
  Morphine consumption

CONTACTS AND LOCATIONS:
Overall Officials: Jing Cang, MD, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China